CLINICAL TRIAL: NCT06358417
Title: CHW Intervention to Improve Nutrition Security of Primary Care Patients With Hypertension
Brief Title: CHW Intervention to Improve Nutrition Security of Patients With Hypertension
Acronym: HeartWell
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Anne N. Thorndike, MD, MPH, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000873
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Nutrition, Healthy; Food Insecurity; Community Health Worker
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition-enhanced CHW intervention (Experimental): This intervention integrates a nutrition component into the Basic CHW hypertension intervention to address gaps in patients' knowledge, skills, and resources for consuming and sustaining a healthful diet. CHWs will administer a 4-part nutrition curriculum that is tailored to the needs and preferences of a food-insecure population with limited resources. The nutrition education materials provided to participants will include a booklet of nutrition information that will serve as the primary educational resource for CHW use with participants.
  Interventions: Behavioral: Nutrition-enhanced CHW
- Basic CHW intervention (Active Comparator): The CHW provides basic hypertension education, coaching about adherence to medications and primary care visits, and home BP cuffs and promotion of BP self-monitoring. All participants are provided home BP cuffs and remote monitoring free of charge.
  Interventions: Behavioral: Basic CHW

INTERVENTIONS:
Behavioral: Nutrition-enhanced CHW — CHW provides nutrition education and skills training in addition to the usual care (Basic CHW) hypertension management.
  Arms: Nutrition-enhanced CHW intervention
Behavioral: Basic CHW — CHW provide usual care for hypertension management.
  Arms: Basic CHW intervention

SUMMARY:
The goal of this study is to implement and evaluate a randomized pilot study of a 4-month Nutrition-enhanced community health worker (CHW) intervention for primary care patients with nutrition insecurity and poorly controlled hypertension. The nutrition intervention will be added to the pre-existing Massachusetts General Hospital CHW hypertension (Basic CHW) program that provides hypertension education, coaching about adherence to medications and primary care visits, and home BP cuffs and promotion of BP self-monitoring over the course of approximately 4 months.

DETAILED DESCRIPTION:
The goal of this study is to implement and evaluate a randomized pilot study of a 4-month Nutrition-enhanced CHW intervention in primary care patients with nutrition insecurity and poorly controlled hypertension. The nutrition intervention will be added to the pre-existing Massachusetts General Hospital CHW hypertension (Basic CHW) that provides basic hypertension education, coaching about adherence to medications and primary care visits, and home BP cuffs and promotion of BP self-monitoring over the course of approximately 4 months. The CHW nutrition intervention curriculum is tailored to the needs and preferences of a food-insecure population with limited resources. Nutrition education materials will be provided to participants, including a booklet of nutrition information and a summarized version of key points on a brochure that they can use as a quick reference when grocery shopping. Nutrition education will focus on reducing sodium, saturated fats, and added sugars and increasing fruits, vegetables, and whole grains. Much of the educational material is based on a traffic-light system. These topics are organized into four modules: nutrition label reading, grocery shopping, meal-planning, and healthy cooking.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to participate in the Massachusetts General Hospital CHW hypertension program (age 21 years or older, uncontrolled hypertension, patient at one of 5 participating primary care clinics; either identifies as a minoritized race/ethnicty or is low-income); speaks English or Spanish

Exclusion Criteria:

* declines participation in CHW hypertension program; does not speak English or Spanish

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasiblity | Baseline
  Proportion of eligible participants enrolled in study
Feasibility of CHW nutrition intervention (intervention arm only) | 4 months
  At least 70% participants complete at least 3 of 4 CHW nutrition education modules
Acceptability (intervention arm only) | 4 months
  Average of participants' ratings of intervention components on a 10-point scale.

SECONDARY OUTCOMES:
Diet quality | 4 months
  Change in Healthy Eating Index-20 score
Blood pressure | 4 months
  Change in systolic and diastolic blood presure
Secondary feasibility (intervention arm only) | 4 months
  At least 70% participants complete 3 of 6 nutrition worksheets
Secondary feasibility (intervention arm only) | 4 months
  At least 70% participants have a CHW assessment of their home cooking environment

CONTACTS AND LOCATIONS:
Overall Officials: Anne N Thorndike, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified feasiblity, acceptability, diet quality, and blood pressure data will be shared. The data and details related to the analytic plan and study measures will be deposited in a publicly accessible data repository, such as the Harvard Dataverse, a NIH-approved Scientific Generalist Data Repository free to researchers inside and outside the Harvard community.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Analytic plans and details will be made available no later than the official publication date of a peer-reviewed article that includes the study results, and these will be available for at least 5 years after the study period ends. De-identified data from the study will be made publicly available through the data repository within 90 days of the closeout of the project and made available according to the Harvard Dataverse's data retention policy.
Access Criteria: In accordance with the data repository methods, completion of a data use agreement form, that stipulates data sharing under an IRB-approved protocol, will be required for accessing the data.

REFERENCES:
- [Derived] Gu KD, Cheng J, Bejarano O, Gelsomin E, Malone A, Faulkner KC, Thorndike AN. Design of Heart Well: A randomized pilot study of a community health worker-delivered nutrition intervention for low-income adults with hypertension. Contemp Clin Trials. 2026 Jan 28;162:108244. doi: 10.1016/j.cct.2026.108244. Online ahead of print. PMID 41610938